CLINICAL TRIAL: NCT07278973
Title: HemoDiafiltration Versus HemoDialysis in OLDER People: a Randomized, Multicenter, Crossover, Pragmatic Clinical Trial
Brief Title: Hemodiafiltration Versus Hemodialysis in Older People
Acronym: HD-OLDER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AUB Santé (Other)
Responsible Party: Principal Investigator, Mabel Aoun, Nephrologist, AUB Santé
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2025-A00884-45
Record Dates: First submitted 2025-09-18; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Hemodialysis; Hemodiafiltration; Fatigue Symptom; Quality of Life of Patients; Older People
Keywords: Hemodialysis; Hemodiafiltration; Older people; Fatigue; Patient reported outcome; Dialysis recovery time
MeSH Terms: conditions — Fatigue | interventions — Hemodiafiltration

STUDY DESIGN:
Masking Description: Data analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1: HD HDF (Experimental): The patient will receive three months of HD followed by three months of HDF
  Interventions: Other: High-flux hemodialysis; Other: Hemodiafiltration
- Sequence 2: HDF HD (Experimental): The patient will receive three months of HDF followed by three months of HD
  Interventions: Other: High-flux hemodialysis; Other: Hemodiafiltration

INTERVENTIONS:
Other: High-flux hemodialysis — High-flux hemodialysis removes small and middle molecular solutes through the mechanism of diffusion.
Other: Hemodiafiltration — Hemodiafiltration removes solutes using convection which allows for more epuration of middle molecular solutes.

SUMMARY:
This study will compare the impact of two hemodialysis techniques on fatigue and post-dialysis recovery time in patients aged 85 years and older. These two techniques are high-flux hemodialysis (HD) and hemodiafiltration (HDF).

Patients will receive the treatment over two periods: if period 1 is HD then period 2 will be HDF. Every patient will be his/her own control, this is why it is called cross-over. Each period will last three months. Between the two periods, patients will receive a traditional low-flux hemodialysis.

These two techniques are widely used worldwide and their side-effects are well-known and do not put the patients at risk. HDF has been shown to improve survival in patients with a mean age of 58 years. But a previous study from the investigators' group showed that HDF causes a prolonged recovery time in older patients. This randomized trial aims to elucidate this question.

DETAILED DESCRIPTION:
Study purpose: To determine the best modality of hemodialysis in older patients > 84 years

Study Design: Randomized, multicenter, crossover, pragmatic clinical trial.

Participants who fulfil the inclusion and exclusion criteria will be randomized in a 1:1 ratio for HDF or high-flux hemodialysis, using the SNOSE method (for allocation concealment).

Patients will be randomized to two sequences, each one of a 3-month period. Sequence 1 includes 3 months of hemodiafiltration (Period 1) then 3 months of high-flux hemodialysis (Period 2). Sequence 2 includes 3 months of high-flux hemodialysis (Period 1) then 3 months of hemodiafiltration (Period 2).

Washout period: Two weeks of low-flux hemodialysis at the beginning of the study and between the two periods of each sequence.

Blinding: the participant, investigators and outcome assessors are not blinded the intervention.

Primary objective: To compare the dialysis recovery time in older patients treated with hemodiafiltration versus conventional high-flux hemodialysis

Secondary objectives

1. To compare the general fatigue between the two hemodialysis modalities
2. To compare symptomatic hypotension and intradialytic clotting events
3. To compare quality of life
4. To compare dialysis adequacy
5. To compare safety and adverse events

Eligibility criteria: described under the section "Eligibility".

Duration of study for each participant: 7 months (including 2 initial weeks of washout and 2 weeks of washout between period 1 and period 2) Total duration of study: 8-10 months

Data collection at screening/randomization

* Eligibility criteria: clearly stated and documented in the eCRF.
* Demographics: age, sex.
* Comorbidities and medical history: diabetes, smoking, hypertension, hyperlipidemia, cause and date of kidney failure (dialysis vintage), previous cardiovascular disease, atrial fibrillation, Charlson score for comorbidity.
* Vital signs: height and weight (dry weight). Pre-dialysis and post-dialysis systolic and diastolic blood pressure and heart rate in a sitting position will be recorded.
* Dialysis prescription: Vascular access (arteriovenous fistula or graft, central venous catheter); number of dialysis hours per week; dialysis session time (morning, afternoon, evening); blood flow, dialysate flow, dialysate temperature, filter membranes (surface), dialysate potassium, sodium, calcium content and type (acetate, HCL or citrate), anticoagulation type and dose (heparin or LMWH) will be collected. Use of UF control (or profile) or Na control (or profile).
* Laboratory pre-dialysis: urea, creatinine, serum phosphate, calcium, albumin, potassium, sodium, bicarbonate, hemoglobin, PTH, alkaline phosphatase, ferritin, transferrin saturation, uric acid, Kt/V (method of Kt/V assessment) to be recorded.
* Laboratory post-dialysis: urea, creatinine.
* Clinical variables: Urine volume will be assessed by collecting the 24 hour-urine and residual kidney function will be measured.
* Medications: antihypertensive therapy: number of drugs, diuretics, renin angiotensin aldosterone system inhibitors (RAASi), CCBs, beta-blockers, alpha-blockers; antidepressants and anxiolytics. Statin, medications for diabetes, oral anticoagulant, ESA, Iron, drugs for hyperkalemia, phosphate binders, vitamin D, cinacalcet.
* Dialysis recovery time (DRT) will be collected for three consecutive sessions and will be assessed by asking "How long did it take you to recover from your last dialysis session?" or in French "Combien de temps vous a-t-il fallu pour récupérer de votre dernière séance d'hémodialyse?". This question will be asked by nurses to each patient at each session for three consecutive sessions at the beginning, middle and end of each period of the trial. Answers will be recorded in minutes or hours.
* Fatigue score will be assessed by using the French SONG-fatigue validated scale. The SONG-HD fatigue scale includes three questions: in the last week, "did you feel tired?", "did you lack energy?", "did fatigue limit your usual activities?". The response to these questions follows a 4-Likert scale: 0= not at all, 1=a little, 2=quite a bit, 3=severely. The total score of fatigue is defined as the sum of the three scores (0 to 9).
* Stand-to-sit (STS 30) test: it is used to evaluate muscle performance and it is validated in patients on hemodialysis. It is assessed by asking the patient at the end of the session for three consecutive sessions to stand and sit on the chair as quickly as possible. The number of stand-to-sit over 30 seconds will be recorded.
* Health-related quality of life will be assessed using the SF-12 quality of life score.

Data collection at follow-up

-Laboratory measurements The investigators will collect at one month, two months and three months of Period 1 and Period 2 the routine laboratory tests: serum urea, creatinine, phosphate, calcium, albumin, potassium, sodium, bicarbonate, hemoglobin, PTH, alkaline phosphatase, ferritin, transferrin saturation.

At the end of each period, residual kidney function will be collected.

* Clinical follow-up: The number of symptomatic intradialytic hypotension episodes and of intradialytic clotting events will be documented in the patient's chart at each session and the total number will be collected at the end of each period of treatment. Pre- and post-dialysis systolic and diastolic blood pressure will be collected at the end of each period of the trial by computing the average of the last three sessions.
* Number of hospital admissions and deaths, within each period, will be collected.
* Dialysis parameters will be collected at one month, two months and three months of each period of the trial: blood flow, dialysate flow, dialysate temperature, ultrafiltration rate (mL/Kg/h), Kt/V, convective volume (for HDF), use of UF control (or profile) or Na control (or profile), dialysis session duration and time (morning, afternoon, evening).
* Medications' follow-up: Any change in baseline medications to be collected every month: antihypertensive therapy, ESA, Iron, drugs for hyperkalemia, phosphate binders, vitamin D, cinacalcet.
* Questionnaires DRT question, SONG-Fatigue questionnaire, STS-30 will be administered and recorded at 6 weeks and the end of Period 1 and Period 2. SF-12 Health Survey will be administered and recorded at the end of Period 1 and Period 2.

Primary and Secondary Endpoints: defined under the section "Outcome measures".

Planned number of participants: 62 patients

Statistical analysis Analyses will be performed on an intention-to-treat basis. Baseline characteristics will be compared using the independent t-test or Mann-Whitney U test for continuous variables and Chi-Square test for categorical variables. Linear mixed models will be used to compare the outcomes.

Ethics: The study will be conducted according to the principles of the Declaration of Helsinki 1975.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Age >84 years
* Diagnosed with kidney failure
* On maintenance hemodialysis >3months
* Willing to have a dialysis session of 3.5 to 4-hour duration, three times a week
* Has a reliable vascular access
* Is covered by the health insurance

Exclusion Criteria:

* Patients with cognitive impairment (assessed with a mini-test if needed)
* Hospitalized at inclusion
* Have difficulties with French speaking
* Terminally ill with life expectancy<3 months
* With active cancer

Min Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12-17 (Estimated); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in dialysis recovery time | Three months
  Time in minutes that the patient needs after dialysis to recover energy

SECONDARY OUTCOMES:
Change in fatigue score | Three months
  Fatigue will be assessed using the Standardized Outcomes in Nephrology (SONG) fatigue scale: from 0 to 9, higher meaning worse outcomes.
Change in STS-30 | Three months
  The number of stand-to-sit over 30 seconds will be recorded. The higher the better outcome.
Change in SF-12 scores | Three months
  Quality of life scale (12 items), from 0 to 100, the higher the better outcome.
Number of episodes of of symptomatic hypotension | Three months
  Drop in blood pressure with symptoms
Number of intradialytic clotting events | Three months
Change in hemoglobin level | Three months
Change in serum albumin | Three months
Change in serum potassium level | Three months
Change in serum phosphate | Three months
Change in Kt/V | Three months
  Dialysis adequacy
Hospitalisation | From the start to the end of period 1 (HD) and from the start to the end of period 2 (HDF)
  Whether the patient was admitted to hospital during the study period
Death | From the start to the end of period 1 (HD) and from the start to the end of period 2 (HDF)

CONTACTS AND LOCATIONS:
Overall Officials: Mabel Aoun, M.D., M.P.H., Study Chair — AUB SANTE
Locations (4):
- France (4):
  - AUB Santé, Bretagne
  - AIDER, Grabels
  - ECHO, Le Mans
  - Aura Paris, Paris

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2025-09-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT07278973/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT07278973/SAP_001.pdf